CLINICAL TRIAL: NCT02548052
Title: A Phase I Trial to Evaluate Safety and Efficacy of Topically Applied GSK2981278 Ointment in a Psoriasis Plaque Test
Brief Title: Study of Safety and Efficacy of Topical GSK2981278 Ointment in Plaque Psoriasis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 201465
Record Dates: First submitted 2015-09-10; First posted 2015-09-14 (Estimated); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Psoriasis
Keywords: retinoic acid receptor-related orphan receptor (ROR) gamma inverse agonist; Plaque type psoriasis; psoriasis plaque test; Topical; GSK2981278
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- GSK2981278, Vehicle, Betamethasone valerate (Experimental): All subjects will receive all six treatments (GSK2981278 ointment 0.03%, 0.1%, 0.8%, 4%, vehicle to match GSK2981278 ointment and betamethasone valerate 0.1% cream); with random assignment of the treatments to 6 test fields on identified stable plaque(s) on the upper extremities, thighs and/or trunk. Subjects will be treated once-daily (except Days 7 and 14) over 19 days (a total of 16 applications) under semi-occlusive conditions (covered by an adhesive non-woven fabric).
  Interventions: Drug: GSK2981278 0.03%; Drug: GSK2981278 0.1%; Drug: GSK2981278 0.8%; Drug: GSK2981278 4%; Drug: Vehicle; Drug: Betamethasone valerate 0.1%

INTERVENTIONS:
Drug: GSK2981278 0.03% — GSK2981278 will be supplied as a white to off-white ointment containing GSK2981278A drug substance at a concentration of 0.03%. Approximately 200 microliters of the GSK2981278 0.03% ointment will be applied topically to the assigned test field once daily.
Drug: GSK2981278 0.1% — GSK2981278 will be supplied as a white to off-white ointment containing GSK2981278A drug substance at a concentration of 0.1%. Approximately 200 microliters of the GSK2981278 0.1% ointment will be applied topically to the assigned test field once daily.
Drug: GSK2981278 0.8% — GSK2981278 will be supplied as a white to off-white ointment containing GSK2981278A drug substance at a concentration of 0.8%. Approximately 200 microliters of the GSK2981278 0.8% ointment will be applied topically to the assigned test field once daily.
Drug: GSK2981278 4% — GSK2981278 will be supplied as a white to off-white ointment containing GSK2981278A drug substance at a concentration of 4%. Approximately 200 microliters of the 4% ointment will be applied topically to the assigned test field once daily.
Drug: Vehicle — GSK2981278 vehicle will be supplied as a white to off-white ointment containing no drug substance. Approximately 200 microliters of the vehicle will be applied topically to the assigned test field once daily.
Drug: Betamethasone valerate 0.1% — Betamethasone valerate will be supplied as a cream. Approximately 200 microliters of the 0.1% betamethasone valerate cream will be applied topically to the assigned test field once daily.

SUMMARY:
GSK2981278 is a highly potent and selective inverse agonist of retinoic acid receptor-related orphan receptor gamma (ROR gamma) that is under development for topical treatment of plaque type psoriasis suitable for topical therapy.

This is the first study to administer GSK2981278 to subjects with psoriasis. This proof-of-concept study will evaluate the safety, tolerability and initial efficacy of a range of concentrations of GSK2981278 ointment with repeated topical applications in adult subjects with psoriasis. Results of this study will provide first clinical information on the drug's safety and efficacy in psoriasis and inform the selection of concentration of GSK2981278 ointment to be evaluated in subsequent clinical studies.

This is a Phase 1, single center, test field-randomized, vehicle- and positive- controlled, subject- and evaluator-blind study. All subjects will receive all 6 treatments on 6 test fields, for intra-individual treatment comparison. For every subject, the manner of assignment of each treatment to a particular test field will be according to a randomization scheme. Thus, the test fields within each subject, and not the subjects themselves, will be randomized.

The study will consist of screening, followed by a treatment period of 19 days, and a follow-up visit at Day 27 (+/-2) for subjects who will consent for biopsy. During the treatment period, subjects will receive all of these treatments: GSK2981278 ointment 0.03% weight by weight [w/w], 0.1% w/w, 0.8% w/w, 4% w/w, GSK2981278 vehicle, and betamethasone valerate 0.1% cream. The test fields on which these treatments will be applied will be identified on stable plaque(s) on the upper extremities, thighs and/or trunk. A blinded evaluator (an investigator or designee) will perform the measurements and assessments whereas an unblinded study staff member (not an evaluator) will perform biopsy collection.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and above, at the time of signing the informed consent.
* Subjects with stable plaque psoriasis for >= 6 months, as confirmed by the subject.
* Up to three plaque area(s) sufficient for six test fields. The target lesion(s) should be on the trunk, upper extremities or thighs (excluding hands and skin folds); psoriatic lesion(s) on the knees or elbows are not to be used as a target lesion. It is recommended, but not required, that all selected plaques are symmetrical in location, size and clinical characteristics.
* Plaques to be treated should have a comparable thickness of the Echo Lucent Band (ELB) (as a surrogate for the psoriatic infiltrate thickness) of at least 200 micrometers on Day 1.
* Male:

Male subjects with female partners of child bearing potential must comply with the following contraception requirements from the time of first dose of study medication until after the last dose of study medication.

1. Vasectomy with documentation of azoospermia.
2. Male condom. These allowed methods of contraception are only effective when used consistently, correctly and in accordance with the product label. The investigator is responsible for ensuring that subjects understand how to properly use these methods of contraception.

   * Female of non-reproductive potential (FNRP):

A FNRP is eligible to participate in this study if she meets at least one of the following conditions:

1. Females with one of the following procedures documented and no plans to utilize assisted reproductive techniques (e.g., in vitro fertilization or donor embryo transfer): Bilateral tubal ligation or salpingectomy; Hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion; Hysterectomy; Bilateral Oophorectomy (surgical menopause)
2. Post-menopausal women (including all women over 60 years of age, see below), Post-Menopause criteria: Females 60 years of age or older; A practical definition accepts menopause after 1 year without menses with an appropriate clinical profile, e.g., age appropriate, >45 years, in the absence of hormone replacement therapy (HRT) or medical suppression of the menstrual cycle (e.g., leuprolide treatment) [In questionable cases for women < 60 years of age, a blood sample with simultaneous follicle stimulating hormone and estradiol falling into the central laboratory's post-menopausal reference range is confirmatory (these levels need to be adjusted for specific laboratories/assays)]; Females under 60 years of age, who are on HRT and wish to continue, and whose menopausal status is in doubt, are required to use a highly effective method to avoid pregnancy, as outlined in the protocol. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrolment. For most forms of HRT, at least 2 to 4 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a highly effective method to avoid pregnancy

   * Capable of giving signed informed consent, which includes compliance with the pre-specified requirements and restrictions.

Exclusion Criteria:

* Alanine aminotransferase (ALT) >2xUpper Limit of Normal (ULN) and bilirubin >1.5x ULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Corrected QT (QTc) interval > 450 milliseconds (msec) or QTc > 480 msec in subjects with Bundle Branch Block. The QTc is the QT interval corrected for heart rate according to Bazett's formula (QTcB), and/or machine-read. The QTc should be based on single QTc values of ECG obtained over a brief recording period.
* Any condition that, in the judgement of the investigator, would put the subject at unacceptable risk for the participation in the trial.
* Current evidence of another ongoing or any acute cutaneous infection, history of repeated or chronic significant skin infections (unless irrelevant in the opinion of the investigator, i.e. onychomycosis, labial herpes or other minor diagnosis).
* Clinically-relevant skin disease, other skin pathologies, or a history of skin cancer, that may, in the opinion of the investigator, contraindicate participation or interfere with test field evaluations.
* History of malignancy within 5 years prior to dosing, except adequately treated noninvasive cancer of the skin (basal or squamous cell).
* Psoriasis other than plaque variants.
* Use of prohibited concomitant medications or products within the defined washout periods before the Day 1 visit and during the trial.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates their participation.
* Contraindications according to summary of product characteristics of the active positive control.
* Symptoms of a clinically significant illness that may, in the opinion of the investigator, influence the outcome of the trial in the 4 weeks before baseline visit and during the trial.
* Presence of hepatitis B surface antigen (HBsAg), positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study treatment.
* A positive pre-study drug/alcohol screen.
* A positive test for human immunodeficiency virus (HIV) antibody.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Prolonged exposure to natural or artificial sources of ultraviolet (UV) radiation within 2 weeks prior to the Day 1 visit or intention to have such exposure during the study, thought by the investigator likely to modify the subject's psoriasis.
* In the opinion of the investigator or physician performing the initial examination the subject should not participate in the clinical trial, e.g. due to probable noncompliance or inability to understand the trial and give adequately informed consent.
* Close affiliation with the investigator (e.g. a close relative) or persons working at Bioskin GmbH or subject is an employee of sponsor.
* Subject is institutionalized because of legal or regulatory order.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-10-22 (Actual); Primary Completion 2016-02-19 (Actual); Study Completion 2016-02-19 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events | From Day 1 until follow-up visit (Day 27)
  An adverse event is any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Change from baseline in clinical laboratory parameters | Baseline and Days 8, 15, and 19
Change from baseline in heart rate | Baseline and Day 19
Change from baseline in systolic and diastolic blood pressure | Baseline and Day 19
Change from baseline in oral temperature | Baseline and Day 19
Change from baseline in electrocardiogram (ECG) | Baseline and Days 15 and 19
  Single 12-lead ECGs will be obtained using an ECG machine that automatically calculates heart rate and measures PR, QRS, QT, and corrected QT (QTc) intervals.
Reduction in infiltrate thickness of the psoriatic plaque(s) from baseline | Baseline (Day 1) and Days 4, 8, 15, and 19
  Infiltrate thickness will be measured by 22-MegaHertz high-frequency sonography. Sonography will be done on Days 1, 4, 8, 15, and 19.

SECONDARY OUTCOMES:
Clinical assessment score using a 5- point scale | Baseline (Day 1) and Days 4, 8, 15, and 19
  Improvement of the test site(s) will be assessed using a 5-point scale with score ranging from -1 (worsened) to 3 (completely healed). Score at Day 1 will be documented as "zero".

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Hamburg, Germany

REFERENCES:
- [Derived] Kang EG, Wu S, Gupta A, von Mackensen YL, Siemetzki H, Freudenberg JM, Wigger-Alberti W, Yamaguchi Y. A phase I randomized controlled trial to evaluate safety and clinical effect of topically applied GSK2981278 ointment in a psoriasis plaque test. Br J Dermatol. 2018 Jun;178(6):1427-1429. doi: 10.1111/bjd.16131. Epub 2018 Mar 23. No abstract available. PMID 29150844
- See also: Results for study 201465 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/201465?search=study&search_terms=201465#rs